CLINICAL TRIAL: NCT07079085
Title: Safety Evaluation of Pueraria Lobata Radix in Specific Consumption Scenarios for Type 2 Diabetes: A Real-World Study
Brief Title: Safety Evaluation of Pueraria Lobata Radix in Specific Consumption Scenarios for Type 2 Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Jiangxi University of Traditional Chinese Medicine (Other)
Collaborators: The Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xu Zhou, Professor, Jiangxi University of Traditional Chinese Medicine
Other Study IDs: JXUCM-DIET-02
Record Dates: First submitted 2025-07-10; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
Keywords: Pueraria lobata radix; Ge Gen; Type 2 diabetes mellitus; Safety; Real-world study
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pueraria lobata radix group: This group includes patients with T2DM who consumed Pueraria lobata radix in any special scenarios.
- Control group: This group includes patients with T2DM who did not consume Pueraria lobata radix in any special scenarios.

SUMMARY:
This real-world study aims to investigate the association between the consumption of Pueraria lobata radix and adverse events in patients with type 2 diabetes mellitus (T2DM) under special scenarios. By retrospectively analyzing the clinical data of patients with T2DM, we will evaluate the safety profile of Pueraria lobata radix in different special populations, identify potential risk factors, and provide evidence-based support for the safe consumption and clinical use of Pueraria lobata radix.

DETAILED DESCRIPTION:
Pueraria lobata radix (PLR), the dried root of Pueraria lobata (Willd.) Ohwi (Family Leguminosae), is an herb with both medicinal and edible applications, historically utilized for treating diabetes. Recent research advances regarding its bioactive constituents have progressively validated PLR's potential efficacy in the adjunctive therapy of type 2 diabetes mellitus (T2DM). Animal studies demonstrate that multiple active compounds within PLR, such as puerarin and polysaccharides, exert significant hypoglycemic effects. The underlying mechanisms include improvement of insulin sensitivity, reduction of insulin resistance, enhancement of glucose tolerance, and protection of pancreatic β-cell function. Based on this evidence, puerarin injections (primarily composed of the standardized extract puerarin) are clinically employed for treating T2DM and its complications, exhibiting substantial therapeutic benefits. Clinical studies further confirm that PLR dietotherapy at conventional doses effectively assists glycemic control with a favorable safety profile. Owing to its dual designation as both a medicine and food, PLR has gained widespread adoption in the daily dietary management of T2DM patients.

However, significant uncertainties persist concerning PLR's safety under non-standard consumption patterns. For instance, some patients may consume PLR products at high doses, for extended durations, or irregularly. Furthermore, consumption occurs among special populations, such as children, pregnant or lactating women, and the elderly. Such usage patterns and dosages may substantially deviate from established recommendations. The absence of systematic safety assessments for these scenarios leaves potential risks unclarified. This safety concern is exacerbated within unregulated market environments; the lack of restrictions on PLR purchase or intake could diminish patient awareness regarding safe dosing practices, thereby elevating risks associated with non-standard use.

To address these gaps, this study will conduct a retrospective real-world investigation to systematically evaluate the safety of PLR under special consumption scenarios within T2DM populations.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis with T2DM.
2. Documented history of consuming Pueraria lobata radix (PLR) in any dosage form (e.g., dried slices, root cubes).
3. Fulfillment of at least one of the following special scenarios: 1) Excessive dosage: Daily PLR intake ≥ twice the maximum dose specified in the Chinese Pharmacopoeia; 2) Long-term consumption: PLR consumption duration ≥ three months with frequency ≥ three times weekly; 3) Advanced age: ≥ 80 years; 4) Pregnancy; 5) Lactation; 6) Allergic constitution: History of any food or drug allergy; 7) Liver dysfunction: Clinical diagnosis of liver cirrhosis or chronic liver failure, or laboratory findings of total bilirubin > 1.5 × upper limit of normal (ULN) or alanine aminotransferase (ALT)/aspartate aminotransferase (AST) > 2 × ULN; 8) Renal insufficiency: Clinical diagnosis of diabetic nephropathy or chronic nephritis with renal function impairment, or serum creatinine > 120% of ULN.
4. Occurrence of adverse events during the retrospective observation period within one month following PLR consumption.

Exclusion Criteria:

1. Diagnosis of type 1 diabetes mellitus, gestational diabetes mellitus, or other specific types of diabetes.
2. Use of PLR compound preparations (e.g., puerarin injection).
3. Unavailability of complete clinical data or patient refusal to provide essential information required for the observation period during follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise individuals diagnosed with T2DM. Diagnosis will be established according to international diabetes guidelines, defined as meeting any of the following criteria: a fasting blood glucose (FBG) level ≥126 mg/dL (7.0 mmol/L), a blood glucose level ≥200 mg/dL (11.1 mmol/L) measured 2 hours after a 75-g oral glucose tolerance test, or a glycated hemoglobin (HbA1c) level ≥6.5% (48 mmol/mol).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of individual adverse events | Collect data from the past 6 months for each sample, with the sample sources spanning a two-year period
  The between-group differences in the incidence of individual adverse events will be compared across the eight predefined special consumption scenarios: 1) excessive dosage, 2) long-term consumption, 3) advanced age, 4) pregnancy, 5) lactation, 6) allergic constitution, 7) liver dysfunction, and 8) renal insufficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhou, M.D, Principal Investigator — Jiangxi University of Traditional Chinese Medicine
Locations (1):
- The Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No